CLINICAL TRIAL: NCT03807973
Title: Tracking Peripheral Immune Cell Infiltration of the Brain in Central Inflammatory Disorders Using [Zr-89]Oxinate-4-labeled Leukocytes.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, MD, PhD, Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R18-179
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome; Multiple Sclerosis; Healthy
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Fibromyalgia (Experimental)
  Interventions: Drug: [Zr-89]Oxine-labeled leukocytes PET/MRI
- Chronic Fatigue Syndrome (Experimental)
  Interventions: Drug: [Zr-89]Oxine-labeled leukocytes PET/MRI
- Multiple Sclerosis (Experimental)
  Interventions: Drug: [Zr-89]Oxine-labeled leukocytes PET/MRI
- Healthy Controls (Experimental)
  Interventions: Drug: [Zr-89]Oxine-labeled leukocytes PET/MRI

INTERVENTIONS:
Drug: [Zr-89]Oxine-labeled leukocytes PET/MRI — All study participants will undergo an investigational imaging study using autologous [Zr-89]-labeled leukocytes and brain PET/MRI. Participants will undergo a venous blood draw, and the leukocytes in the blood sample will be isolated for labeling using [Zr-89]oxine. The labeled leukocytes (7.4- 18.5 megabecquerel (MBq), 200-500 uCi) will be re-injected into the participant followed by brain PET/MRI at 24-48 hours after injection. Participants will be asked to have a second brain imaging study 3-6 days after this injection, but this second imaging study is optional.

SUMMARY:
This study will use brain Positron Emission Tomography/ Magnetic Resonance Imaging (PET/MRI) and an investigational radioactive drug called [Zr-89]oxine to track the location of white blood cells (also called leukocytes) in the body. PET/MRI will be used to visualize labeled white blood cells and determine if they enter the central nervous system in conditions associated with brain inflammation (also called neuroinflammation). By better understanding the role of neuroinflammation in fibromyalgia, chronic fatigue syndrome, and multiple sclerosis, the investigator hopes to be able to better diagnose and treat patients in the future.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 65 years of age 2.Healthy volunteer OR

* Clinical diagnosis of Multiple Sclerosis (MS) OR
* Meets 2016 American College of Rheumatology (ACR) case definition criteria for fibromyalgia OR
* Meets 1994 Fukuda case definition criteria for Chronic Fatigue Syndrome

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy
3. Lactation
4. Individuals who are unable to participate in the imaging portion due to severity of their medical condition
5. Chronic infectious disease (e.g. HIV, HCV)
6. Viral or bacterial illness requiring medical attention and/or antibiotics within 1 month of study participation
7. Diagnosis of cancer, including leukemia
8. Blood or blood clotting disorder
9. Except for individuals with MS, a diagnosis of autoimmune disease is exclusionary
10. Positive urine pregnancy test day of procedure or a serum pregnancy test within 48 hours prior to the administration of Zirconium-89 Oxinate-4-labeled leukocytes
11. Currently enrolled in a clinical trial utilizing experimental therapies
12. Contraindication to gadolinium based contrast agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Regional brain distribution of radiolabeled white blood cells | 3 years
  Descriptive statistics (means and standard deviations) of standardized uptake values (SUVs) will be presented for the patient groups and healthy controls in the following regions: whole brain, gray matter, white matter, atlas-based regions of interest, and lesions (MS patients only). Normality of the SUV distribution will be tested using Shapiro-Wilk tests, and the data will be transformed to normal distribution if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD,PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States